CLINICAL TRIAL: NCT05008510
Title: Phase 2 Clinical Efficacy and Safety Study of Sabizabulin (VERU-111) Monotherapy and Sacituzumab Govitecan-hziy/Sabizabulin Combination Therapy for the Treatment of Metastatic Triple Negative Breast Cancer
Brief Title: P2 Clinical Efficacy & Safety Study of V-111 Monotherapy & Sacituzumab Govitecan-hziy/V-111 Combo Therapy for mTNBC .
Acronym: VERU-111
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided to halt and will potentially reopen in the future.
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V2011801
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Metastatic Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sabizabulin

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, randomized, open-label, three treatment-arm, efficacy and safety study. Subjects will be randomized to the three treatment arms.
Who Masked: Outcomes Assessor
Masking Description: Central reader for scans will be blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sabizabulin Monotherapy (Experimental): Subjects in the Sabizabulin Treated Group will receive sabizabulin 32 mg each day by mouth until disease progression confirmed by BICR is observed.
  Interventions: Drug: Sabizabulin
- Sacituzumab govitecan-hziy/Sabizabulin Combination (Experimental): Subjects in the Sacituzumab govitecan-hziy /Sabizabulin Combination Treated Group will receive sabizabulin 32 mg each day by mouth and Sacituzumab govitecan-hziy at the FDA approved dose and dosage regimen for mTNBC until disease progression confirmed by BICR is observed.
  Interventions: Drug: Sabizabulin/Sacituzumab govitecan-hziy Combo
- Sacituzumab govitecan-hziy Monotherpy (Active Comparator): Subjects in the Control Treated Group will receive Sacituzumab govitecan-hziy intravenous infusion of 10 mg/kg in accordance with the FDA approved use and dosage regimen for mTNBC until disease progression confirmed by BICR is observed.
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sabizabulin — Sabizabulin (Veru-111)
  Other Names: Veru-111
  Arms: Sabizabulin Monotherapy
Drug: Sacituzumab Govitecan-hziy — Sacituzumab govitecan-hziy
  Arms: Sacituzumab govitecan-hziy Monotherpy
Drug: Sabizabulin/Sacituzumab govitecan-hziy Combo — Sabizabulin/Sacituzumab govitecan-hziy Combo therpy
  Other Names: Sacituzumab govitecan-hziy and Veru-111 combo
  Arms: Sacituzumab govitecan-hziy/Sabizabulin Combination

SUMMARY:
To compare the following:

1. The efficacy of sabizabulin monotherapy to sacituzumab govitecan-hziy monotherapy
2. The efficacy of sacituzumab govitecan-hziy/sabizabulin combination therapy to sacituzumab govitecan-hziy monotherapy

These comparisons will be made in the efficacy in the treatment of metastatic triple negative breast cancer (mTNBC) in patients previously treated with at least two systemic chemotherapies for metastatic disease as measured by radiographic progression free survival (rPFS) as the primary endpoint.

DETAILED DESCRIPTION:
Stage 1: This is a safety run-in portion of the study for the combination therapy. Three subjects will be enrolled into Stage 1 of the study to receive sacituzumab govitecan-hziy for injection + sabizabulin 32 mg. Dosing with sabizabulin should be within 1 hour prior to initiation of the sacituzumab govitecan-hziy infusion.

Safety will be assessed for 21 days. Samples for assessment of pharmacokinetics of sacutizumab (in the Control Treated Group and TS Combination Group), and sabizabulin (in the Sabizabulin Treated Group and TS Combination Group) will be collected on Day 1 (prior to dosing and within 1 hour after the sacituzumab govitecan-hziy infusion has been completed in Stage 1 and Stage 2, Cycle 1 only), Day 3 (prior to dosing with sabizabulin, Stage 1, Cycle 1 only), and Day 8 (prior to dosing and within 1 hour after the sacituzumab govitecan-hziy infusion has been completed in Stage 1 and Stage 2, Cycle 1 only).

The primary objective of Stage 1 is to demonstrate an acceptable safety profile of the combination therapy regimen that is planned for Stage 2 of the protocol. If an acceptable safety profile and no unacceptable drug related adverse event is observed in Stage 1, then Stage 2 will be initiated as designed. If an unacceptable drug related adverse event is observed in one patient in the combination treatment group in Stage 1, then an additional 3 patients will be enrolled to the combination treatment arm. If 2 out of 3 or 2 out of 6 patients experience an unacceptable drug related adverse event in Stage 1, then the combination treatment regimen will not be dosed in Stage 2 of this protocol.

Stage 2: This study is a multicenter, randomized, open-label, three treatment-arm, efficacy and safety study. Subjects will be randomized to the three treatment arms.

Patients will be randomized in a 1:1:1 fashion to the sacituzumab govitecan-hziy monotherapy, sabizabulin monotherapy, and the sacituzumab govitecan-hziy/sabizabulin combination therapy treatment arms.

Subjects in the Sabizabulin Treated Group and sacituzumab govitecan-hziy/sabizabulin Combination Group will receive sabizabulin 32 mg per day orally until radiographic progression (blinded independent central read) in observed. Subjects in the Control Treated Group and in the sacituzumab govitecan-hziy/sabizabulin Combination Group will receive sacituzumab govitecan-hziy using the dose and dosing regimen defined in the FDA approved prescribing information for the treatment of mTNBC until radiographic progression in observed.

The primary efficacy endpoint of the study will be the median rPFS. Subjects will continue study treatment until disease progression confirmed by blinded independent central reader (BICR) is observed. A follow up visit will occur approximately 30 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Be able to communicate effectively with the study personnel
* Aged ≥18 years
* For Female Subjects
* Menopausal status Be postmenopausal as defined by the National Comprehensive Cancer

Network as either:

* Age ≥55 years and one year or more of amenorrhea
* Age <55 years and one year or more of amenorrhea, with an estradiol assay <20 pg/mL
* Age <55 years and surgical menopause with bilateral oophorectomy Be premenopausal or perimenopausal with a negative urine pregnancy test. If subject is of child-bearing potential, the subject must agree to use acceptable methods of contraception:
* If female study participant could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization of male partner (vasectomy with documentation of azoospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}
* If female study participant has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used
* If female study participant has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used
* For Male Subjects
* Subject must agree to use acceptable methods of contraception:

If the study subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e., barrier method of contraception], surgical sterilization (vasectomy with documentation of azoospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)

* If female partner of a study subject has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used
* If female partner of a study subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used
* If female partner of a study subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS), a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Histologically or cytologically confirmed TNBC based on the most recent analyzed biopsy or other pathology specimen. Triple negative defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PR) and negative for human epidermal growth factor receptor 2 (HER2) by in-situ hybridization.
* Measurable disease is required as per RECIST 1.1 confirmed by BICR (NOTE: Bone only metastatic disease is acceptable but requires a measurable component).
* Refractory to or relapsed after at least two prior standard chemotherapy regimens for advanced/metastatic TNBC and have not received Sacituzumab govitecan-hziy.
* At least 2 weeks beyond prior anti-cancer treatment (chemotherapy, radiotherapy, and/or major surgery), and recovered from all acute toxicities to Grade 1 or less (except alopecia and peripheral neuropathy).
* At least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids < 20 mg prednisone or equivalent daily are permitted).
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, ANC > 1,500 per mm3, platelets > 100,000 per mm3).
* Adverse events at study entry < Grade 1 by NCI CTCAE v5.0 (Patients with ≤ Grade 2 neuropathy and any grade of alopecia are eligible).
* Patients with treated, non-progressive brain metastases, off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks can be enrolled in the trial.
* Subject is willing to comply with the requirements of the protocol through the end of the study.

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential or fertile men with a female partner of childbearing potential not willing to use effective contraction during the study and 6 months after last dose of study drug for the women of childbearing potential participating in the study and for 3 months after last dose of study drug in fertile men with a female partner of childbearing potential.
* Known hypersensitivity or allergy to sabizabulin or Sacituzumab govitecan-hziy
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 X upper limit of normal (ULN) or total bilirubin >ULN (an elevated total bilirubin up to 1.5 X ULN attributed to a previously confirmed diagnosis of Gilbert's disease is acceptable if all other eligibility criteria are met). In patients with documented metastases to the liver, the limits for inclusion are ALT or AST >5.0 X ULN or total bilirubin >1.5 X ULN.
* Patients with biliary catheter
* Creatinine Clearance ≤60 mL/min by the Cockroft-Gault equation
* Has a known additional, invasive, malignancy that is progressing or required active treatment in the last 5 years (note: subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or cervical carcinoma in situ that have undergone potentially curative therapy are not excluded)
* Any comorbid disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Infection requiring antibiotic use within one week or randomization or uncontrolled infection.
* Treatment with any investigational product within < 4 half-lives for each individual investigational product OR within 28 days prior to randomization
* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or within 60 days after the final dose of study treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of sabizabulin monotherapy to Sacituzumab govitecan-hziy monotherapy | 360 days
  The comparison will be made in the efficacy in the treatment of metastatic triple negative breast cancer (mTNBC) in patients previously treated with at least two systemic chemotherapies for metastatic disease as measured by radiographic progression free survival (rPFS) as the primary endpoint.
To compare the efficacy of Sacituzumab govitecan-hziy/sabizabulin combination therapy to Sacituzumab govitecan-hziy monotherapy | 360 days
  The comparison will be made in the efficacy in the treatment of metastatic triple negative breast cancer (mTNBC) in patients previously treated with at least two systemic chemotherapies for metastatic disease as measured by radiographic progression free survival (rPFS) as the primary endpoint.

SECONDARY OUTCOMES:
Objective Response Rate (ORR), proportion of subjects with a best tumor response of ORR (PR or CR) on study | 360 days
  Objective Response Rate (ORR), proportion of subjects with a best tumor response of ORR (PR or CR) on study

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.

IPD SHARING:
Plan to Share IPD: Undecided